CLINICAL TRIAL: NCT04009174
Title: Multi-modality Prostate Cancer Image Guided Interventions
Acronym: IGPC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101038
Record Dates: First submitted 2018-10-24; First posted 2019-07-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PET/CT; PET/MRI; Fluorocholine; PSMA; Sodium (Na) MRI; [18-F]-FCH; [18-F]-DCFPyL; Hybrid imaging; Whole mount histopathology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging Panel (Experimental): Patients who provided written informed consent and found to be eligible for study were asked to complete Positron Emission Tomography (PET) + Dynamic CT imaging, PET/MRI (with endorectal coil) and 3D-Transrectal ultrasound prior to standard of care radical prostatectomy.
  Interventions: Other: Imaging Panel

INTERVENTIONS:
Other: Imaging Panel — Initial Protocol (REB approval date 08-Sept-2011)
  Pre-operative Imaging Panel
  * [18F]-FCH PET + Dynamic CT
  * MRI of the pelvis with endorectal coil (T1, T2, DW, DCE, MRS)
  * 3D-Transrectal ultrasound
  * Optional PET/MRI (added with Protocol Amend 1, REB approval date 22-Aug-2012)
  * Optional Sodium (23Na) MRI (added with Protocol Amend 2, REB approval date 25-Feb-2013)
  Protocol Amendment #3, REB approval date 20-Oct-2015:
  Pre-operative Imaging Panel
  * [18-F]-DCFPyL PET+Dynamic CT
  * PET/MRI with endorectal coil
  * 3D-Transrectal Ultrasound
  * Optional Sodium (23Na) MRI

SUMMARY:
This is a non-randomized, prospective trial of men who are scheduled for radical prostatectomy for treatment of prostate cancer, or repeat biopsy for localized prostate cancer as standard of care and who will undergo a series of pre-operative multi-modality imaging studies. Post intervention, hybrid imaging maps (HIM) will be generated and the predictions of the HIM (3D location, volume and grade of cancer) will be correlated with actual pathology results to gauge the performance of the HIM in both radical prostatectomy and biopsy settings.

DETAILED DESCRIPTION:
This study was built on our first study (IGPC-1, REB number 15551) which acquired multi-modality imaging in 36 patients undergoing radical prostatectomy. We successfully demonstrated the ability to accurately co-register pre-operative multi-modality images (MRI: T1, T2, Diffusion Weighed (DW), Dynamic Contrast enhanced (DCE); Dynamic Contrast Enhanced CT, 3D Ultrasound with post-operative whole mount pathology specimens. We have developed a platform for the segmentation of prostate cancer on the whole mount pathology specimens and are in the process of analyzing the data to develop a hybrid imaging map (HIM) of prostate cancer distribution (location and grade) based on the correlation of the pre-operative imaging signals and the post-operative pathology (citation provided below). The HIM will need subsequent validation in a separate cohort of radical prostatectomy patients and evaluated as to its ability to be incorporated as a targeting tool for prostate interventions such as prostate biopsy and this is the purpose of this follow-up study.

On the IGPC-2 study, pre-operative imaging panels were successfully obtained in 24 patients accrued to cohort 1. The protocol was then amended to include [18-F]-DCFPyl instead of [18F]-FCH. [18-F]-DCFPyl was a newer PET probe that may possess superior performance because it is directed against prostate specific membrane antigen (PSMA), a protein commonly expressed on prostate cancer cells. Imaging-pathology correlations in the first 6 patients imaged with [18-F]-DCFPyl were compared to the correlations obtained with [18F]-FCH imaging in the first 24 patients.

IGPC-2 Cohort 1 (Radical Prostatectomy) was expanded to provide an additional 20 men imaged with [18-F]-DCFPyl as part of the imaging panel. The goal was to acquire 24 complete imaging datasets with [18-F]-DCFPyl as the PET imaging agent to enable us to draw comparisons with the 24 [18F]-FCH imaging data sets acquired.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent for this study
* Male, aged 18 years or older
* Pathologically confirmed prostate cancer on previous biopsy
* Suitable for and consenting to Radical Prostatectomy for treatment, or repeat biopsy as standard of care

Exclusion Criteria:

* Prior therapy for prostate cancer (including hormone therapy), with the exception of radiation therapy for Cohort 2 only
* Use of 5-alpha reductase inhibitors, i.e. finasteride (Proscar) or dutasteride (Avodart) within 6 months of study start. Patients undergoing a 6-month washout period prior to study start will be eligible.
* Inability to comply with the pre-operative imaging panel
* Patients scheduled for radical prostatectomy with prostate size exceeding dimensions for whole mount pathology slides
* Allergy to contrast agents to be used as part of the imaging panel
* Sickle cell disease or other anemias
* Insufficient renal function (eGFR < 60 mL/min/1.73 m2)
* Residual bladder volume > 150 cc (determined by post-void ultrasound)
* Hip prosthesis, vascular grafting that is MRI incompatible or sources of artifact within the pelvis
* Contraindication to MRI

  * pacemaker or other electronic implants
  * known metal in the orbit
  * cerebral aneurysm clips

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with a prostate
Enrollment: 52 (Actual)
Dates: Start 2012-02-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Hybrid Imaging Map (HIM) Validation | Within two years of study completion.
  We will determine if individualized hybrid imaging maps (HIMs) based on a pre-operative imaging panel accurately predicts the actual cancer distribution found in the whole mount prostatectomy specimens obtained from the surgery.

OTHER OUTCOMES:
MRI Prostate Sodium Imaging Validation | Within two years of study completion
  We will determine if sodium levels in the prostate based on a pre-operative sodium MRI accurately predicts the actual cancer distribution found in the whole mount prostatectomy specimens obtained from the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Glenn Bauman, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymized study data such as de-identified images, digital pathology slides, prostate tissue slides and prostate cancer diagnosis information can be available for data analysis.
Access Criteria: Institutionally approved material sharing agreement.

REFERENCES:
- [Background] Ward A, Crukley C, McKenzie C, Montreuil J, Gibson E, Gomez JA, et al. Registration of in vivo prostate magnetic resonance images to digital histopathology images. MICCAI'10 Proceedings of the 2010 international conference on Prostate cancer imaging: computer-aided diagnosis, prognosis, and intervention; Bejing, China. Berlin: Springer-Verlag; 2010.
- [Derived] Yang DM, Alfano R, Bauman G, Thiessen JD, Chin J, Pautler S, Moussa M, Gomez JA, Rachinsky I, Gaed M, Chung KJ, Ward A, Lee TY. Short-duration dynamic [18F]DCFPyL PET and CT perfusion imaging to localize dominant intraprostatic lesions in prostate cancer: validation against digital histopathology and comparison to [18F]DCFPyL PET/MR at 120 minutes. EJNMMI Res. 2021 Oct 15;11(1):107. doi: 10.1186/s13550-021-00844-0. PMID 34652551
- [Derived] Yang DM, Li F, Bauman G, Chin J, Pautler S, Moussa M, Rachinsky I, Valliant J, Lee TY. Kinetic analysis of dominant intraprostatic lesion of prostate cancer using quantitative dynamic [18F]DCFPyL-PET: comparison to [18F]fluorocholine-PET. EJNMMI Res. 2021 Jan 4;11(1):2. doi: 10.1186/s13550-020-00735-w. PMID 33394284